CLINICAL TRIAL: NCT07387380
Title: KIRA Uterine Drain Device Evaluation - First-In- Human Study
Brief Title: KIRA Uterine Drain Device Evaluation- First-In- Human Study
Acronym: RANI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lucie Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CP-01
Record Dates: First submitted 2026-01-06; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Delivery Procedures
Keywords: cesarean delivery; surgical drain; blood loss measurement
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Interventional (Experimental): All participants will be assigned to the interventional arm, in which the uterine drain is used to evaluate the blood loss immediately following cesarean delivery.
  Interventions: Device: Uterine drain for use in cesarean section

INTERVENTIONS:
Device: Uterine drain for use in cesarean section — The intervention will be used to remove uterine contents and measure blood loss immediately following cesarean delivery.

SUMMARY:
The purpose of this research is to evaluate a new investigational medical device, the Kira device, intended to make it easier for the surgical team to monitor blood loss during and immediately after cesarean deliveries (c-sections). This study will assess the safety of the device and the device's ability to gently suction blood from the uterus into a clear container where it can be seen and measured by the surgical team.

ELIGIBILITY:
Inclusion Criteria:

* Adult, sex female at birth, age 18 years or older at the time of consent.
* Able to understand and provide informed consent to participate in the study.
* Undergoing c-section

Exclusion Criteria:

* Ongoing intrauterine pregnancy
* Untreated uterine rupture
* Unresolved uterine inversion
* Known uterine, cervical, or vaginal anomaly that would prohibit device placement.
* Placenta abnormality including a) known placenta accreta, b) retained placenta with known risk factors for placenta accreta (e.g. history of prior uterine surgery, including prior c-section and placenta previa), c) retained placenta without easy manual removal.
* Diagnosis of coagulopathy
* Current cervical cancer
* Current purulent infection of vagina, cervix or uterus.
* History of allergy to device materials (thermoplastic elastomers (TPE), acrylonitirile butadiene styrene plastic (ABS), cyanoacrylate)
* Lack of study consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and seriousness of device related Adverse Events (ADE's) | Measured at study exit, approximately 3 days

SECONDARY OUTCOMES:
Ease of use questionnaire | Within 2 weeks of study completion
  Likert type scale with higher scores indicating agreement with the statement.
Cumulative blood loss | Measured through 24 hours from time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study for a commercial product.